CLINICAL TRIAL: NCT01906190
Title: Persistence Study of Immune Response After Vaccination With Influenza Vaccine in Healthy Population
Brief Title: Persistence of Immune Response After Vaccination With Influenza Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Principal Investigator, Wu Jiang, Department of Immunization & Prevention, Beijing Centers for Disease Control and Prevention, Centers for Disease Control and Prevention, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BJCDCWJ201104
Record Dates: First submitted 2013-07-09; First posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Influenza, Human; Immunisation Reaction
Keywords: influenza vaccine; immune response; persistence
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vaccinated group (Experimental): Vaccinated group means that subjects whose antibodies less than 1:40 6 months later after primary vaccination will receive a booster dose of seasonal influenza vaccine.
  Interventions: Biological: seasonal influenza vaccine

INTERVENTIONS:
Biological: seasonal influenza vaccine — subjects whose antibodies less than 1:40 6 months later after primary vaccination will receive a booster dose of seasonal influenza vaccine

SUMMARY:
This clinical study will be performed in subjects aged 12-60 years old enrolled in NCT01310374 who received 2010 seasonal influenza vaccine to evaluate the persistence of the immune response of influenza vaccine up to 24 months after vaccination.

DETAILED DESCRIPTION:
Subjects were previously vaccinated at 12 to 60 years of age with 2010 seasonal influenza vaccine.The persistence phase starts 24 months after the primary vaccination and blood samples will be taken at 6, 12, 18 and 24 months after primary vaccination. Subjects whose antibody titer less than 1:40 at 6 months after primary vaccination will receive a booster dose of influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* aged 12-60 years old
* male or non-pregnant female
* volunteers received 2010 seasonal influenza vaccine
* clinically healthy as determined by: medical history inquiring and physical examination
* provide written informed consents before joining the trial

Exclusion Criteria:

* without history of 2010 seasonal influenza vaccine administration,
* allergic to any ingredient of vaccine,
* autoimmune disease or immunodeficiency,
* severe adverse reaction after vaccination, such as allergies, hives, breathing difficulties, angioedema or abdominal pain,
* severe acute and chronic diseases
* axillary temperature over 37.0℃ at the time of vaccination.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 207 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
change from serum antibodies against vaccine-related influenza virus at 6,12,18,24 months | 6，12，18，24 months after the primary vaccination
  Persistence of antibodies in all subjects with respect to components of the investigational vaccine - month 6，12，18，24

CONTACTS AND LOCATIONS:
Overall Officials: jiang wu, Bachelor, Principal Investigator — Beijing Centers for Disease Control and Prevention
Locations (1):
- Tuoketuo Centers for Disease Control & Prevention, Tuoketuo County, Inner Mongolia, China